CLINICAL TRIAL: NCT00816010
Title: A Multicentre, Randomised Study to Examine the Effects of Telephone Intervention in Patients With Coronary Heart Disease and Diabetes
Brief Title: Telephone Intervention in Patients With Acute Coronary Syndrome (ACS) and Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of manpower at the various study sites
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Wing-Yee So, Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Telephone intervention
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus; Acute Coronary Syndrome
Keywords: drug compliance; lifestyle modification
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Acute Coronary Syndrome; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lifestyle and compliance counseling via telephone contact with structured set of questions and reinforcements provided
  Interventions: Behavioral: telephone contact
- 2 (No Intervention): Control arm with usual care as per local hospital practice

INTERVENTIONS:
Behavioral: telephone contact — for lifestyle and compliance counseling
  Arms: 1

SUMMARY:
Hypothesis To investigate whether telephone counselling by nurse educator between clinic visits with particular emphasis on adherence to medications and lifestyle modification in patients with coronary heart disease and diabetes will reduce mortality and hospitalisation rates due to cardiovascular events compared to usual clinic-based care.

DETAILED DESCRIPTION:
Study-design A 2-year multicentre, randomised controlled open study involving 5 HA hospitals in Hong Kong.

Subjects and method One thousand two hundred and sixteen patients admitted to hospital with principle diagnosis of coronary heart disease and known or newly confirmed diabetes on oral glucose tolerance test will be enrolled. Patients in the intervention arm (n=608) will receive telephone intervention between clinic visits by diabetes nurse educator using structured counselling tools with particular emphasis on adherence to lifestyle modification and medications as well as self-monitoring of blood glucose, blood pressure and body weight. Patients in control group (n=608) will not receive telephone intervention. Both groups will be followed up by their usual medical teams in their hospitals upon discharge.

Clinical endpoints Primary endpoint is the composite of death and/or cardiovascular related hospitalisations. Secondary endpoints include hospitalisations due to cardiovascular events, number of hospital admissions, total number of days of hospital stay and attendance at the Accident and Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the 5 HA hospitals with principle diagnosis of CHD, age 45 years for male and 55 for female
* Presence of diabetes according to the 1998 WHO criteria and no history of unprovoked ketosis and not requiring continuous insulin treatment within 1 year of diagnosis

Exclusion Criteria:

* Patients with terminal malignancy or other life-threatening diseases with less than 3-month expected survival
* Telephone contact not available
* Patients with a mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Patients who speak non-Cantonese dialect or different language or have conditions that prevent effective communications e.g. patients who are deaf and mute
* Patients who live in nursing home with supervised treatment
* Patients who have participated in another intervention study during the last 1 month and who are enrolled in any intervention studies.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of death and/or CVD related hospitalisations (acute myocardial infarction, revascularisation procedures, heart failure or unstable angina or arrhythmia requiring hospital admissions, lower extremity amputation and stroke) by 24 months. | 24 months

SECONDARY OUTCOMES:
Cardiovascular endpoints | 24 months
Number of hospital admissions, total number of days of hospitalization | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wing Yee So, MRCP, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- 5 public hospitals in Hong Kong, Hong Kong, Hong Kong